CLINICAL TRIAL: NCT01155791
Title: A Phase I Study Evaluating the Efficacy and Safety of Sodium Selenite in Combination With Docetaxel in Castration-resistant Prostate Cancer
Brief Title: Phase I Sodium Selenite in Combination With Docetaxel in Castration-resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Sandy Srinivas (Other)
Responsible Party: Sponsor-Investigator, Sandy Srinivas, Associate Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROS0033; SU-05122010-6002 (Other: Stanford University); 17356 (Other: Stanford IRB)
Record Dates: First submitted 2010-06-30; First posted 2010-07-02 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Urologic Neoplasms; Prostate Cancer; Prostate Cancer Metastatic Disease
MeSH Terms: conditions — Urologic Neoplasms; Prostatic Neoplasms | interventions — Docetaxel; Prednisone

ARMS (1):
- combination sodium selenite and docetaxel (Experimental)
  Interventions: Drug: Docetaxel; Drug: Biosyn; Drug: Prednisone

INTERVENTIONS:
Drug: Docetaxel — IV 75 mg/m2
Drug: Biosyn — IV dosage varies
Drug: Prednisone — 5mg, orally

SUMMARY:
Selenium, in the form of inorganic Sodium Selenite, may be useful for treating existing prostate cancer. This idea is based on data from our laboratory showing that 1) prostate cancer cells are more sensitive to Selenium (Sodium Selenite)-induced apoptosis than normal prostate epithelial cells, 2) Selenite induces significant growth inhibition of well established prostate cancer tumors in mice at doses that have no detectable toxicity, and 3) Selenite disrupts AR signaling, and that the inhibition of AR expression and activity by Selenite occurs via a redox mechanism involving GSH, superoxide, and Sp1. Altogether, these findings suggest that Selenium may be useful in a variety of potential indications in the natural history of prostate cancer, including both hormone sensitive and castrate resistant prostate cancer, as a single agent, or in combination with radiation, chemotherapy or conventional hormone therapy. Selenite is a potential novel inhibitor of AR expression and function in prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate
2. Castration-resistant prostate cancer requires the following 3 criteria:

   * Failure of first line bilateral orchiectomy or therapy with an LHRH agonist,
   * A rising PSA on 3 consecutive occasions at least 1 week apart (but not limited to the 30 day screening period), AND
   * A castrate level of testosterone (<50ng/dL)
3. PSA doubling time (PSADT) > 1 months
4. Failure on docetaxel chemotherapy as defined by a rising PSA .
5. A minimum PSA of 2 ng/mL
6. Age >=18 years
7. Life expectancy greater than 6 months
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 or Karnofsky performance status >=80%
9. Bone metastases will be allowed
10. The subject has a QTcB (Bazett corrected) or QTcF (Frederica corrected) < 470 msec.
11. Ability to understand and the willingness to sign a written informed consent document.
12. Willingness to stay on docetaxel chemotherapy despite rising PSA level.

Exclusion Criteria:1. Radiotherapy for prostate cancer within 28 days prior to Day 1.

2. More than 1 prior chemotherapy

3. Inadequate organ function, as evidenced by any of the following at screening:

* Absolute neutrophil count (ANC) < 1500/uL
* Platelet count <= 100 x 10^9/L
* Total bilirubin >= ULN
* AST, and/or ALT > 1.5 x the upper limit of normal (ULN) with a concomitant alkaline phosphastase >2.5 X ULN
* Serum creatinine > 2.0 mg/dL
* Hemoglobin < 9 g/dL

  4. Men with reproductive potential who do not agree to use an accepted and effective method of contraception during the study treatment period and for at least 3 months after completion of the study treatment.

  5. History of other malignancies within 5 years prior to Day 1 except for tumors with a negligible risk for metastasis or death, such as adequately controlled basal cell carcinoma, squamous-cell carcinoma of the skin, or early-stage bladder cancer

  6. Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study.

  7. Known or prior treated brain metastases.

  8. History of hypersensitivity to docetaxel

  9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure ,unstable angina pectoris, cardiac arrhythmia, significant vascular disease (e.g. aortic aneurysm, aortic dissection), symptomatic peripheral vascular disease, or psychiatric illness/social situations that would limit compliance with study requirements.

  10. History of myocardial infarction or unstable angina within 6 months prior to study enrollment

  11. History of stroke or transient ischemic attack within 6 months prior to study enrollment 12. The subject is known to be positive for the human immunodeficiency virus (HIV) and is receiving antiretroviral 12. Willingness to stay on docetaxel chemotherapy despite rising PSA level.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of the combination sodium selenite and docetaxel after 4 cycles of combination therapy using the NCI Common Toxicity Criteria v3.0 grading system for adverse events | after 4 cycles of combination therapy
To determine the maximum tolerated dose (MTD) | 1 cycle

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sandy Srinivas, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States